CLINICAL TRIAL: NCT04446910
Title: Using Technology to Reduce Youth Substance Use
Acronym: TEXT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1K24DA046569-01A1 (NIH); 1K24DA046569-01A1 (NIH)
Record Dates: First submitted 2020-05-07; First posted 2020-06-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Drug Use
Keywords: Adolescent; Juvenile justice; text messaging; Substance use; mHealth
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a hybrid 1 effectiveness-implementation design in which the investigators will test a theory-driven digital health (i.e., SMS text-messaging) treatment engagement intervention while also collecting data on the text messaging platform's potential implementation and adoption within juvenile justice and behavioral health settings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS Text Messaging (Experimental): SMS text messaging intervention for a period of 90 days to encourage attendance at community-based substance use or dual diagnosis treatment appointments through motivational messages.
  Interventions: Behavioral: SMS Text Messaging
- Standard of Care Engagement Practices (Active Comparator): Standard of care engagement practices, such as communicating with youth and caregivers, as needed, through texting but frequency of contact and content of messaging varies according to individual needs.
  Interventions: Behavioral: Standard of Care Engagement Practices

INTERVENTIONS:
Behavioral: SMS Text Messaging — SMS text messaging intervention for a period of 90 days to promote attendance at community-based substance use or dual diagnosis treatment appointments through motivational messages.
  Arms: SMS Text Messaging
Behavioral: Standard of Care Engagement Practices — Standard of care engagement practices, such as communicating with youth and caregivers, as needed, through texting but frequency of contact and content of messaging varies according to individual needs.
  Arms: Standard of Care Engagement Practices

SUMMARY:
The research project will focus on conducting a trial of whether a tailored SMS text-messaging intervention is efficacious in improving justice-involved youths' substance use or dual diagnosis treatment attendance and engagement.

DETAILED DESCRIPTION:
The study will demonstrate how delivery of motivational/coaching messages to justice-involved youth and their caregivers will lead to greater youth substance use treatment attendance and engagement. The study will start with identifying the feasibility and acceptability of the SMS text-messaging intervention with community-supervised justice-involved youth. Then, the study will determine whether the tailored dyadic (youth and caregiver) SMS text-messaging intervention improves justice-involved youth substance use or dual diagnosis treatment attendance and engagement relative to standard of care (not receiving motivational/coaching messages). Finally, the study will characterize patterns of key justice and behavioral health system-level factors that promote or hinder eventual adoption and sustainability of mHealth technology as a tool to improve treatment attendance for justice-involved youth.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking youth with willing adult caregiver
* Ages 13-18
* Justice-involved while living in the community
* Own a mobile phone or tablet
* Are willing to send and receive text messages
* Are referred to community-based substance use and/or mental health treatment

Exclusion Criteria:

-

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Treatment session attendance | 30 days post baseline
  Proportion of treatment sessions attended
Treatment session attendance | 60 days post baseline
  Proportion of treatment sessions attended
Treatment session attendance | 90 days post baseline
  Proportion of treatment sessions attended
Treatment session attendance | 120 days post baseline
  Proportion of treatment sessions attended
Treatment session attendance | 180 days post baseline
  Proportion of treatment sessions attended

SECONDARY OUTCOMES:
First treatment session initiation | 120 days post baseline
  Proportion who attended first treatment session, as scheduled
First treatment session initiation | 180 days post baseline
  Proportion who attended first treatment session, as scheduled

OTHER OUTCOMES:
Alcohol use | 90 days post baseline
  The Adolescent Risk Behavior Assessment (ARBA) is used to assess quantity and frequency of previous (lifetime and past 90 days) alcohol use.
Alcohol use | 180 days post baseline
  The Adolescent Risk Behavior Assessment (ARBA) is used to assess quantity and frequency of previous (lifetime and past 90 days) alcohol use.
Drug use | 90 days post baseline
  The Adolescent Risk Behavior Assessment (ARBA) is used to assess quantity and frequency of previous (lifetime and past 90 days) cannabis and other drug use.
Drug use | 180 days post baseline
  The Adolescent Risk Behavior Assessment (ARBA) is used to assess quantity and frequency of previous (lifetime and past 90 days) cannabis and other drug use.
Drug Use | 90 days post baseline
  The Texas Christian University (TCU) Drug Screen with Opioid Supplement is used to gather detailed information about drug and opioid use.
Drug Use | 180 days post baseline
  The Texas Christian University (TCU) Drug Screen with Opioid Supplement is used to gather detailed information about drug and opioid use.
Response rate to SMS messages | 30 days post baseline
  Digital (mobile) health metrics
Response rate to SMS messages | 60 days post baseline
  Digital (mobile) health metrics
Response rate to SMS messages | 90 days post baseline
  Digital (mobile) health metrics
Psychiatric symptoms | 90 days post baseline
  Global Appraisal of Individual Needs-Short Screener (GAIN-SS) is used to identify people with recent and lifetime internalizing and externalizing mental health disorders, substance use disorders and crime/violence problems. GAIN-SS responses are given in terms of the recency of the problem described in the questions: 3 = past month; 2 = 2 to 12 months ago; 1 = 1+ years ago; 0 = never. The number of past-month symptoms (number of 3s) is used as a measure of change; the number of past-year symptoms (number of 3s or 2s) is used to identify who is likely to have a current diagnosis; and the number of lifetime symptoms (number of 3s, 2s, or 1s) is used as a covariate measure of lifetime severity.
Psychiatric symptoms | 180 days post baseline
  Global Appraisal of Individual Needs-Short Screener (GAIN-SS) is used to identify people with recent and lifetime internalizing and externalizing mental health disorders, substance use disorders and crime/violence problems. GAIN-SS responses are given in terms of the recency of the problem described in the questions: 3 = past month; 2 = 2 to 12 months ago; 1 = 1+ years ago; 0 = never. The number of past-month symptoms (number of 3s) is used as a measure of change; the number of past-year symptoms (number of 3s or 2s) is used to identify who is likely to have a current diagnosis; and the number of lifetime symptoms (number of 3s, 2s, or 1s) is used as a covariate measure of lifetime severity.
Therapeutic Alliance | 30 days post baseline
  The Working Alliance Inventory (WAI) is used to assess youth's perception of therapeutic alliance (with treatment provider) over time. Scores range from 12 to 84 with higher scores indicating greater perceived therapeutic alliance.
Therapeutic Alliance | 60 days post baseline
  The Working Alliance Inventory (WAI) is used to assess youth's perception of therapeutic alliance (with treatment provider) over time. Scores range from 12 to 84 with higher scores indicating greater perceived therapeutic alliance.
Therapeutic Alliance | 90 days post baseline
  The Working Alliance Inventory (WAI) is used to assess youth's perception of therapeutic alliance (with treatment provider) over time. Scores range from 12 to 84 with higher scores indicating greater perceived therapeutic alliance.
Therapeutic Alliance | 120 days post baseline
  The Working Alliance Inventory (WAI) is used to assess youth's perception of therapeutic alliance (with treatment provider) over time. Scores range from 12 to 84 with higher scores indicating greater perceived therapeutic alliance.
Therapeutic Alliance | 180 days post baseline
  The Working Alliance Inventory (WAI) is used to assess youth's perception of therapeutic alliance (with treatment provider) over time. Scores range from 12 to 84 with higher scores indicating greater perceived therapeutic alliance.
Treatment Motivation | 30 days post baseline
  The Motivation for Youth's Treatment Scale (MYTS) is used to measure intrinsic treatment motivation.
Treatment Motivation | 60 days post baseline
  The Motivation for Youth's Treatment Scale (MYTS) is used to measure intrinsic treatment motivation.
Treatment Motivation | 90 days post baseline
  The Motivation for Youth's Treatment Scale (MYTS) is used to measure intrinsic treatment motivation.
Treatment Motivation | 120 days post baseline
  The Motivation for Youth's Treatment Scale (MYTS) is used to measure intrinsic treatment motivation.
Treatment Motivation | 180 days post baseline
  The Motivation for Youth's Treatment Scale (MYTS) is used to measure intrinsic treatment motivation.
Characteristics of Communication and Interaction with Probation Officers and Treatment Providers | 30 days post baseline
  Questions on communication characteristics will identify the preferred modes and patterns of communication between caregivers/youth and probation officers/treatment providers.
Characteristics of Communication and Interaction with Probation Officers and Treatment Providers | 60 days post baseline
  Questions on communication characteristics will identify the preferred modes and patterns of communication between caregivers/youth and probation officers/treatment providers.
Characteristics of Communication and Interaction with Probation Officers and Treatment Providers | 90 days post baseline
  Questions on communication characteristics will identify the preferred modes and patterns of communication between caregivers/youth and probation officers/treatment providers.
Characteristics of Communication and Interaction with Probation Officers and Treatment Providers | 120 days post baseline
  Questions on communication characteristics will identify the preferred modes and patterns of communication between caregivers/youth and probation officers/treatment providers.
Characteristics of Communication and Interaction with Probation Officers and Treatment Providers | 180 days post baseline
  Questions on communication characteristics will identify the preferred modes and patterns of communication between caregivers/youth and probation officers/treatment providers.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Tolou-Shams, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No